CLINICAL TRIAL: NCT01416415
Title: Glaucoma Eye Drop Instillation: Impact of Education
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not practical to continue due interim results
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Angelo Tanna, Vice Chairman, Department of Ophthalmology and Director, Glaucoma Service, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NU 00051931
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Glaucoma, Open-Angle
Keywords: Glaucoma, Open-Angle; Ophthalmic Solutions, Eye drops; Instructional Films and Videos
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational intervention (Experimental): The educational intervention arm will contain subjects who will watch a video on proper eye drop instillation technique.
  Interventions: Other: Video education on proper eye drop instillation technique
- Attention placebo (Placebo Comparator): The attention control placebo group will receive an educational intervention that mimics the amount of time and attention received by the treatment group. The video chosen is regarding healthy eating tips.
  Interventions: Other: Placebo video education on healthy eating tips

INTERVENTIONS:
Other: Video education on proper eye drop instillation technique — The video is approximately seven minutes long and teaches the Robert Ritch method of instilling eye drops.
  Arms: Educational intervention
Other: Placebo video education on healthy eating tips — The video is approximately seven minutes long and teaches tips to promote healthy eating.
  Arms: Attention placebo

SUMMARY:
The purpose of this study is to assess whether an educational intervention will have a positive effect on patients' ability to properly administer eye drops. The investigators predict that the educational intervention will have a positive impact on the efficacy, safety, and efficiency with which patients administer their eye drops.

DETAILED DESCRIPTION:
Glaucoma is a leading cause of irreversible vision loss worldwide, and as such has a large public health impact. The only treatment proven to slow or arrest the progression of the disease process is intraocular pressure (IOP) reduction, which relies heavily on patient cooperation. Previously, nonadherence to glaucoma medications has ranged from 24% to 59%. Barriers to medication compliance in the glaucoma patient population include health literacy, poor comprehension of disease, poor comprehension of medication regimen, and improper eye drop administration technique. The purpose of this randomized, controlled clinical trial is to assess whether an educational intervention will have a positive effect on patients' ability to properly administer eye drops. Patients randomized to the experimental group will receive the educational intervention, consisting of an instructional video demonstrating how to instill eyedrops. Patients randomized to the control group will receive an attention placebo, consisting of a video regarding healthy eating tips. Additional measures that will be obtained from all patients include a health literacy score, as measured using the REALM questionnaire, and a BMQ - specific score (Beliefs about Medicines Questionnaire) using the BMQ-specific questionnaire. If the education protocol is found to positively affect eye drop administration success, as demonstrated by a statistically significant difference between the experimental and control groups, suggestions will be proposed for the implementation of educational programs similar to ours to improve glaucoma patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Established care with the treating ophthalmologist for at least 6 months
* Diagnosis of open-angle glaucoma or ocular hypertension
* The use of one, two or three self-instilled eye drop medications in one or two eyes
* Age 40-85 years
* Fluency in English
* Best corrected visual acuity (BCVA) of 20/50 or better in each eye

Exclusion Criteria:

* Presence of moderate to severe cognitive deficits
* Presence of a clinically significant tremor
* Mini Mental Status Exam score ≤ 20

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Eye drop instillation score | 4 +/- 3 months
  The eye drop instillation score is a composite score of the efficacy, safety, and efficiency with which the subject instills their eyedrops and is simply a measure of how well the subject administers their eyedrops.

CONTACTS AND LOCATIONS:
Overall Officials: Angelo P Tanna, M.D., Principal Investigator — Northwestern University Department of Ophthalmology
Locations (1):
- Northwestern Medical Faculty Foundation, Chicago, Illinois, United States

REFERENCES:
- [Background] Kulkarni SV, Damji KF, Buys YM. Medical management of primary open-angle glaucoma: Best practices associated with enhanced patient compliance and persistency. Patient Prefer Adherence. 2008 Feb 2;2:303-14. doi: 10.2147/ppa.s4163. PMID 19920977
- [Background] Nemesure B, Honkanen R, Hennis A, Wu SY, Leske MC; Barbados Eye Studies Group. Incident open-angle glaucoma and intraocular pressure. Ophthalmology. 2007 Oct;114(10):1810-5. doi: 10.1016/j.ophtha.2007.04.003. Epub 2007 Jun 20. PMID 17583352
- [Background] The Advanced Glaucoma Intervention Study (AGIS): 7. The relationship between control of intraocular pressure and visual field deterioration.The AGIS Investigators. Am J Ophthalmol. 2000 Oct;130(4):429-40. doi: 10.1016/s0002-9394(00)00538-9. PMID 11024415
- [Background] Kass MA, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Gordon MO. The Ocular Hypertension Treatment Study: a randomized trial determines that topical ocular hypotensive medication delays or prevents the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):701-13; discussion 829-30. doi: 10.1001/archopht.120.6.701. PMID 12049574
- [Background] The effectiveness of intraocular pressure reduction in the treatment of normal-tension glaucoma. Collaborative Normal-Tension Glaucoma Study Group. Am J Ophthalmol. 1998 Oct;126(4):498-505. doi: 10.1016/s0002-9394(98)00272-4. PMID 9780094
- [Background] Lichter PR, Musch DC, Gillespie BW, Guire KE, Janz NK, Wren PA, Mills RP; CIGTS Study Group. Interim clinical outcomes in the Collaborative Initial Glaucoma Treatment Study comparing initial treatment randomized to medications or surgery. Ophthalmology. 2001 Nov;108(11):1943-53. doi: 10.1016/s0161-6420(01)00873-9. PMID 11713061
- [Background] Gold DT, McClung B. Approaches to patient education: emphasizing the long-term value of compliance and persistence. Am J Med. 2006 Apr;119(4 Suppl 1):S32-7. doi: 10.1016/j.amjmed.2005.12.021. PMID 16563940
- [Background] Vakil N. Increasing compliance with long-term therapy: avoiding complications and adverse events. Rev Gastroenterol Disord. 2005;5 Suppl 2:S12-7. PMID 16369223
- [Background] Gurwitz JH, Glynn RJ, Monane M, Everitt DE, Gilden D, Smith N, Avorn J. Treatment for glaucoma: adherence by the elderly. Am J Public Health. 1993 May;83(5):711-6. doi: 10.2105/ajph.83.5.711. PMID 8484454
- [Background] Schwartz GF. Compliance and persistency in glaucoma follow-up treatment. Curr Opin Ophthalmol. 2005 Apr;16(2):114-21. doi: 10.1097/01.icu.0000156139.05323.26. PMID 15744142
- [Background] Tsai JC, McClure CA, Ramos SE, Schlundt DG, Pichert JW. Compliance barriers in glaucoma: a systematic classification. J Glaucoma. 2003 Oct;12(5):393-8. doi: 10.1097/00061198-200310000-00001. PMID 14520147
- [Background] Rotchford AP, Murphy KM. Compliance with timolol treatment in glaucoma. Eye (Lond). 1998;12 ( Pt 2):234-6. doi: 10.1038/eye.1998.56. PMID 9683946
- [Background] Patel SC, Spaeth GL. Compliance in patients prescribed eyedrops for glaucoma. Ophthalmic Surg. 1995 May-Jun;26(3):233-6. PMID 7651690
- [Background] Dietlein TS, Jordan JF, Luke C, Schild A, Dinslage S, Krieglstein GK. Self-application of single-use eyedrop containers in an elderly population: comparisons with standard eyedrop bottle and with younger patients. Acta Ophthalmol. 2008 Dec;86(8):856-9. doi: 10.1111/j.1755-3768.2007.01155.x. Epub 2008 May 20. PMID 18494743
- [Background] Djafari F, Lesk MR, Harasymowycz PJ, Desjardins D, Lachaine J. Determinants of adherence to glaucoma medical therapy in a long-term patient population. J Glaucoma. 2009 Mar;18(3):238-43. doi: 10.1097/IJG.0b013e3181815421. PMID 19295380
- [Background] Gelb L, Friedman DS, Quigley HA, Lyon DW, Tan J, Kim EE, Zimmerman TJ, Hahn SR. Physician beliefs and behaviors related to glaucoma treatment adherence: the Glaucoma Adherence and Persistency Study. J Glaucoma. 2008 Dec;17(8):690-8. doi: 10.1097/IJG.0b013e31816b3001. PMID 19092468
- [Background] Friedman DS, Hahn SR, Quigley HA, Kotak S, Kim E, Onofrey M, Eagan C, Mardekian J. Doctor-patient communication in glaucoma care: analysis of videotaped encounters in community-based office practice. Ophthalmology. 2009 Dec;116(12):2277-85.e1-3. doi: 10.1016/j.ophtha.2009.04.052. Epub 2009 Sep 10. PMID 19744715